CLINICAL TRIAL: NCT00069680
Title: Genetic Analysis of Gray Platelet Syndrome
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030313; 03-HG-0313
Record Dates: First submitted 2003-09-29; First posted 2003-09-30 (Estimated); Last update posted 2018-10-22 (Actual); Status verified 2018-05-17

CONDITIONS: Genetic Linkage; Myelofibrosis
Keywords: Gene Identification; Linkage Analysis; Homozygosity Mapping; Gray Platelet Syndrome; GPS; Platelet Function Defect; Bleeding Disorder
MeSH Terms: conditions — Primary Myelofibrosis; Gray Platelet Syndrome; Hemostatic Disorders

SUMMARY:
This study will identify and characterize the gene or genes responsible for Gray Platelet syndrome (GPS). Platelets are small blood cells that stick on injured blood vessels to form a plug and stop bleeding. When a blood vessel is injured (like a cut on a finger), platelets release the proteins stored in their sacs to help form a blood clot. Patients with GPS bleed longer than other people because their platelets lack some of these protein-carrying sacs. Platelets without sacs look pale gray under the microscope rather than pink, giving the syndrome its name. Except for rare patients with severe hemorrhage, the bleeding tendency in GPS is usually mild to moderate, with patients experiencing easy bruising, nosebleeds, and, in women, excessive menstrual bleeding.

Patients with GPS and members of their family with GPS may be eligible for this study. Participants will provide a personal and family medical history and will have blood drawn. About 1 to 2 tablespoons of blood will be drawn in adults, and about 1 teaspoon in children. The blood will be analyzed for genes that cause GPS

DETAILED DESCRIPTION:
Patients with Gray Platelet Syndrome (GPS) and their unaffected family members will be studied to identify the gene(s) involved in GPS using linkage analysis and gene mapping strategies. Up to 200 individual members of GPS families will be investigated to identify candidate regions of the human genome, which will be further studied using fine mapping and sequence analysis. Characterization of gene(s) involved in GPS could provide important insight into the mechanisms of vesicle formation and protein sorting in human cells.

ELIGIBILITY:
* INCLUSION CRITERIA:

Enrollment in this study will be limited to patients diagnosed with GPS and their unaffected relatives. The diagnosis will be based upon absence or marked reduction of platelet Alpha-granules on electron microscopy.

EXCLUSION CRITERIA:

Patients with reduction in both Alpha and Beta granules will be excluded, since this is probably a separate disease.

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2003-09-29; Study Completion 2018-05-17

CONTACTS AND LOCATIONS:
Overall Officials: Meral Gunay-Aygun, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Raccuglia G. Gray platelet syndrome. A variety of qualitative platelet disorder. Am J Med. 1971 Dec;51(6):818-28. doi: 10.1016/0002-9343(71)90311-1. No abstract available. PMID 5129551
- [Background] White JG. Ultrastructural studies of the gray platelet syndrome. Am J Pathol. 1979 May;95(2):445-62. PMID 453324
- [Background] Levy-Toledano S, Caen JP, Breton-Gorius J, Rendu F, Cywiner-Golenzer C, Dupuy E, Legrand Y, Maclouf J. Gray platelet syndrome: alpha-granule deficiency. Its influence on platelet function. J Lab Clin Med. 1981 Dec;98(6):831-48. PMID 6458643
- [Derived] Gunay-Aygun M, Zivony-Elboum Y, Gumruk F, Geiger D, Cetin M, Khayat M, Kleta R, Kfir N, Anikster Y, Chezar J, Arcos-Burgos M, Shalata A, Stanescu H, Manaster J, Arat M, Edwards H, Freiberg AS, Hart PS, Riney LC, Patzel K, Tanpaiboon P, Markello T, Huizing M, Maric I, Horne M, Kehrel BE, Jurk K, Hansen NF, Cherukuri PF, Jones M, Cruz P, Mullikin JC, Nurden A, White JG, Gahl WA, Falik-Zaccai T. Gray platelet syndrome: natural history of a large patient cohort and locus assignment to chromosome 3p. Blood. 2010 Dec 2;116(23):4990-5001. doi: 10.1182/blood-2010-05-286534. Epub 2010 Aug 13. PMID 20709904